CLINICAL TRIAL: NCT01086280
Title: Comparison of Risk of Major Cardiovascular Events Between Patients With Type 2 Diabetes Initiating Saxagliptin and Those Initiating Other Oral Antidiabetic Treatments
Brief Title: Risk of Cardiovascular Events in Patients With Type 2 Diabetes Initiating Oral Antidiabetic Treatments
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CV181-099
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed to Saxagliptin
- Patients exposed to oral antidiabetic drugs (not Saxagliptin)

SUMMARY:
The purpose of this study is to compare the incidence of major cardiovascular events among patients with type 2 diabetes who are new initiators of Saxagliptin and those who are new initiators of oral anti-diabetic drugs (OADs)in classes other than Dipeptidyl peptidase IV (DPP4) inhibitors.

DETAILED DESCRIPTION:
Prospectively designed retrospective database study. This study will be conducted using administrative claims data and electronic medical records that are collected as part of routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly prescribed Saxagliptin or an OAD in a class other than DPP4 inhibitors
* Enrolled in the respective database for at least 180 days prior to the first prescription for Saxagliptin or other OAD in a class other than DPP4 inhibitors

Exclusion Criteria:

* Patients identified with a diagnostic code for any of the cardiovascular outcomes of interest within the 180-day baseline period
* Patients prescribed a DPP4 inhibitor during the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out using databases containing administrative claims data (HIRD and Medicare in the U.S.) and electronic medical records (GPRD and THIN in the UK). The US population includes patients from health plans in the northeast, southeastern, mid-Atlantic, central, mid-western, and western regions (HIRD) as well as US citizens 65 years of age and older (Medicare). The UK population includes patients seeking medical care from general practitioners (GPRD and THIN)
Sampling Method: Non-Probability Sample
Enrollment: 113505 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events defined as a composite of acute MI, stroke or death due to acute MI, stroke, CHF, dysrhythmia, sudden death, or coronary revascularization. Alternative outcomes include DVT, PE, and arterial vascular disease | 18-months
  Myocardial infarction (MI), congestive heart failure (CHF), deep venous thrombosis (DVT), pulmonary embolism (PE)
Major cardiovascular events defined as a composite of acute MI, stroke or death due to acute MI, stroke, CHF, dysrhythmia, sudden death, or coronary revascularization. Alternative outcomes include DVT, PE, and arterial vascular disease | 36-months
Major cardiovascular events defined as a composite of acute MI, stroke or death due to acute MI, stroke, CHF, dysrhythmia, sudden death, or coronary revascularization. Alternative outcomes include DVT, PE, and arterial vascular disease | 54-months

SECONDARY OUTCOMES:
Acute MI, acute stroke, death from cardiovascular causes, and coronary and carotid revascularization procedures, evaluated separately and then combined | 18-months
Acute MI, acute stroke, death from cardiovascular causes, and coronary and carotid revascularization procedures, evaluated separately and then combined | 36-months
Acute MI, acute stroke, death from cardiovascular causes, and coronary and carotid revascularization procedures, evaluated separately and then combined | 54-months
All-cause death | 18-months
All-cause death | 36-months
All-cause death | 54-months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Lo Re V, Carbonari DM, Saine ME, Newcomb CW, Roy JA, Liu Q, Wu Q, Cardillo S, Haynes K, Kimmel SE, Reese PP, Margolis DJ, Apter AJ, Reddy KR, Hennessy S, Bhullar H, Gallagher AM, Esposito DB, Strom BL. Postauthorization safety study of the DPP-4 inhibitor saxagliptin: a large-scale multinational family of cohort studies of five outcomes. BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000400. doi: 10.1136/bmjdrc-2017-000400. eCollection 2017. PMID 28878934
- [Derived] Saine ME, Carbonari DM, Newcomb CW, Nezamzadeh MS, Haynes K, Roy JA, Cardillo S, Hennessy S, Holick CN, Esposito DB, Gallagher AM, Bhullar H, Strom BL, Lo Re V 3rd. Determinants of saxagliptin use among patients with type 2 diabetes mellitus treated with oral anti-diabetic drugs. BMC Pharmacol Toxicol. 2015 Apr 2;16:8. doi: 10.1186/s40360-015-0007-z. PMID 25889498
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4452&filename=Cv181_099.pdf